CLINICAL TRIAL: NCT02272322
Title: Transvaginal Treatment of Symptomatic Cystocele Grade II-III Using Cousin Biomesh Soft Prolaps or Allium Medical Endofast Reliant
Brief Title: Transvaginal Treatment of Symptomatic Cystocele Grade II-III
Acronym: BCR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Slabbaert Koen (Other)
Responsible Party: Sponsor-Investigator, Slabbaert Koen, MD, Regionaal Ziekenhuis Heilig Hart Tienen
Organization: Regionaal Ziekenhuis Heilig Hart Tienen (Other)
Other Study IDs: BCR-11-01
Record Dates: First submitted 2014-10-01; First posted 2014-10-22 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Cystocele
Keywords: Anterior prolapse
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: cystocele repair with biomesh soft prolaps and endofast reliant

SUMMARY:
This observational study will evaluate treatment of symptomatic cystocele grade II-III with Cousin Biomesh and Allium Medical Endofast Reliant. Data about 100 patients will be collected. Follow-up till 3 years after the procedure. Primary endpoint is absence of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a woman
* Patient is between 40 and 90 years old
* Patient has to sign the informed consent form prior to the procedure
* Patient has to agree with the scheduled follow-up visits on month 1, month 6, year 1, year 2 and year 3
* Patient has symptomatic anterior prolapse

Exclusion Criteria:

* Recurrence cystocele
* Patient is pregnant
* Patient has a wish to become pregnant
* Patient is taking Plavix, Sintrom, Marcoumar, Marevan, Brilique, Efient, Ticlid, Xarelto, Eliquis or Pradaxa. If intake is stopped prior to procedure, patient is allowed to be included.
* Patient is taking LMWH in a dose of more than 40 mg/day
* Patient has a life expectancy < 1 year
* Patient has a known connective tissue disease
* Patient has a history of surgery of the anterior vaginal wall or pelvis
* A scheduled hysterectomy during the index-procedure

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic anterior prolapse
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Absence of recurrence | 3 years

SECONDARY OUTCOMES:
Technical success | day 1
  Correct positioning of the mesh as intended by the surgeon
Procedural success | 30 days
  Technical success without complications till 30 days after the index-procedure
Peroperative complications | day 1
  Perforation bowels, bladder or arteries
Postoperative complications | 3 years
  Infection, bleeding, recurrence, mesh erosion, pain during sexual activities, pain, discomfort
Quality of life | 3 years
  PFDI-20, PFIQ-7, PISQ-12

CONTACTS AND LOCATIONS:
Overall Officials: Koen Slabbaert, MD, Principal Investigator — RZ Heilig Hart Tienen
Locations (1):
- RZ Heilig Hart Tienen, Tienen, Vlaams-Brabant, Belgium